CLINICAL TRIAL: NCT03706508
Title: Pentafecta Outcomes After Robot-assisted Laparoscopic Radical Prostatectomy: First 120 Cases in Brazilian University Hospital
Brief Title: Pentafecta Outcomes After Robot-assisted Laparoscopic Radical Prostatectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Other Study IDs: 2016/0457
Record Dates: First submitted 2018-10-11; First posted 2018-10-16 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-09

CONDITIONS: Prostate Cancer; Erectile Dysfunction; Complication of Surgical Procedure; Urinary Incontinence
Keywords: Robot-assisted prostatectomy; Pentafecta; Biochemical failure; Surgical margin
MeSH Terms: conditions — Prostatic Neoplasms; Erectile Dysfunction; Urinary Incontinence; Margins of Excision

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Robot-assisted laparoscopic radical prostatectomy — Patients with localized prostate cancer underwent transperitoneal robot-assisted laparoscopic radical prostatectomy

SUMMARY:
Robot-assisted laparoscopic radical prostatectomy (RALRP) is a surgical technique for the treatment of prostate cancer. The aim of this study was to report our initial experience with RALRP, by applying the concept of pentafecta. Pentafecta consists of the five main outcomes in the postoperative period of RALRP: erectile dysfunction, urinary incontinence, postoperative complications, surgical margins and biochemical failure.

DETAILED DESCRIPTION:
This study will describe a initial experience in RALRP in Brazilian University Hospital. The follow-up of patients was performed as an examination at the medical consultation every three months. Complications were categorized according to the Clavien classification system. Biochemical failure was established by PSA level. Continence was defined as patients who remain dry and who do not require any kind of protection in their everyday activities. Sexual potency was defined as the ability to get and keep an erection for long enough to have satisfying sexual relations with or without the use of type-5 phosphodiesterase inhibitors (PDE-5) and a Sexual Health Inventory for Men (SHIM) score greater or equal to 21. Positive surgical margin is defined as the presence of neoplastic glands in direct contact with the ink on the surface of the piece, with no interposed connective tissue.

ELIGIBILITY:
Inclusion Criteria:

• patients diagnosed with localized Prostate Adenocarcinoma submitted to surgical treatment with Robot-assisted laparoscopic radical prostatectomy

Exclusion Criteria:

* patients undergoing other treatments for adenocarcinoma of the prostate
* conversion to open prostatectomy
* loss of follow-up

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients between 40 and 75 diagnosed with localized prostate cancer submitted to robot-assisted laparoscopic radical prostatectomy.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2013-08-09 (Actual); Primary Completion 2018-11-30 (Estimated); Study Completion 2018-11-30 (Estimated)

PRIMARY OUTCOMES:
Erectile Dysfunction | 6 months
  Sexual Health Inventory for Men (SHIM) score greater or equal to 21.

SECONDARY OUTCOMES:
Urinary Continence | 6 months
  Continence was defined as patients who remain dry and who do not require any kind of protection.Patients will be questioned in the postoperative consultations if there is a need to use some protection.
Surgical Complication | 30 days
  Complications were categorized according to the Clavien classification system.
Biochemical Failure | 6 month
  Biochemical failure was established by PSA level grater or equal to 0,2 ng/ml.
Surgical Margin | 15 days
  It is defined as the presence of neoplastic glands in direct contact with the ink on the surface of the piece.

CONTACTS AND LOCATIONS:
Overall Officials: Brasil S Neto, PhD, Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided